CLINICAL TRIAL: NCT00004688
Title: Phase II Study of Carmustine, Streptozocin, and Mercaptopurine for Refractory or Recurrent Brain Neoplasms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/13310; EUSM-FDR001274
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-03

CONDITIONS: Anaplastic Astrocytoma; Anaplastic Oligodendroglioma; Mixed Gliomas; Glioblastoma Multiforme; Recurrent Brain Tumor
Keywords: adult anaplastic astrocytoma; adult anaplastic oligodendroglioma; adult brain stem glioma; adult brain tumor; adult glioblastoma multiforme; adult infiltrating astrocytoma; brain tumor; genetic condition; miscellaneous sites/terms; mixed gliomas; nervous tissue tumors; oncologic disorders; rare disease; recurrent adult brain tumor
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma; Glioma; Glioblastoma; Brain Neoplasms; Genetic Diseases, Inborn; Rare Diseases | interventions — Carmustine; Mercaptopurine; Streptozocin

INTERVENTIONS:
Drug: carmustine
Drug: mercaptopurine
Drug: streptozocin

SUMMARY:
OBJECTIVES:

I. Assess the clinical response of patients with refractory or recurrent brain neoplasms treated with carmustine, streptozocin, and mercaptopurine.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive mercaptopurine IV on days 1-3, carmustine by continuous infusion on days 3-5, and streptozocin IV over 20 minutes on days 2-5. Patients receive treatment every 42 days, for up to 4 courses.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Histologically proven refractory or recurrent brain neoplasms Glioblastoma multiforme Anaplastic astrocytoma Gliosarcoma Anaplastic oligodendroglioma Mixed anaplastic glioma Unequivocally progressive primary brainstem tumors following primary therapy Measurable disease --Prior/Concurrent Therapy-- Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior chemotherapy At least 6 weeks since prior nitrosoureas or mitomycin Endocrine therapy: Not specified Radiotherapy: Prior radiotherapy allowed Surgery: Prior surgery allowed --Patient Characteristics-- Age: Not specified Performance status: ECOG 0-2 Karnofsky 60-100% Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT no greater than 4 times normal Renal: Creatinine no greater than 2.0 mg/dL Pulmonary: FEV1 greater than 1 L if symptomatic pulmonary disease present Other: No other concurrent malignancies Not pregnant or lactating Negative pregnancy test Fertile patients must use effective contraception

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35
Dates: Start 1996-08; Study Completion 1998-07

CONTACTS AND LOCATIONS:
Overall Officials: Mark R. Gilbert, Study Chair — Emory University